CLINICAL TRIAL: NCT02930434
Title: Effects of Antarctic Environment on Vitamin D Status and Health Risk Biomarkers of Its Inhabitants
Acronym: AntarD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fuerza Aérea de Chile (Other Government); Instituto Antártico Chileno (Unknown); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-148; RT_28-15 (Other: Instituto Antártico Chileno)
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; cholecalciferol; Antarctica; Chile; cathelicidin; bone metabolism; cardiovascular risk
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard daily vitamin D3 (Active Comparator): Cholecalciferol 600 IU daily during one year or exit from Antarctica.
  Interventions: Dietary Supplement: cholecalciferol
- Higher weekly vitamin D3 (Active Comparator): Cholecalciferol 25000 IU once weekly during one year or exit from Antarctica.
  Interventions: Dietary Supplement: cholecalciferol

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Administration of vitamin D3
  Other Names: Vitamin D3

SUMMARY:
The purpose of this study is to evaluate vitamin D (VD) deficiency in the population of Chilean Antarctica and evaluate the efficacy and safety of VD supplementation to decrease VD deficiency and favorably influence biomarkers for bone, cardiovascular, and immune health risk in the inhabitants of Chilean Antarctica.

DETAILED DESCRIPTION:
The present study consists of an initial cross-sectional evaluation of VD status and specific health biomarkers in inhabitants of Chilean Antarctica, followed by a randomized controlled trial evaluating two acceptable approaches of vitamin D supplementation (cholecalciferol 600 IU daily vs. 25000 IU weekly) in Antarctic inhabitants.

ELIGIBILITY:
Inclusion Criteria:

* population of all ages living in the Chilean Antarctic territory during at least 3 months.

Exclusion Criteria:

* acute or chronic renal disease
* hyper or hypocalcemia
* osteomalacia or Paget's disease of bone
* use of VD supplements or fish oil supplements in the past month in doses higher than 400 IU daily
* treatment for known VD deficiency in the last 6 months
* UV phototherapy in the past month.

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12-10 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Change in serum 25-hydroxyvitamin D concentration | at end of Antarctic residency or 1 year (90-365 days), whichever came first
  In Antarctic inhabitants not supplemented with VD that exit Antarctica before start of RCT phase of study.

SECONDARY OUTCOMES:
sun exposure | at 0, 6, 12 months of Antarctic residency
  questionnaires
sleep pattern | at 0, 6, 12 months of Antarctic residency
  questionnaires
food intake of VD | at 0, 6, 12 months of Antarctic residency
  Food frequency questionnaire
serum biomarkers for bone metabolism | at baseline and every 3 months during supplementation (3,6,9,12 months) up to end of Antarctic residency or 1 year (90-365 days), whichever came first
  intact PTH, calcium phosphorus, alkaline phosphatases, VD-binding protein
serum high-sensitivity C-reactive protein (hsCRP) | at baseline and every 3 months during supplementation (3,6,9,12 months) up to end of Antarctic residency or 1 year (90-365 days), whichever came first
serum cathelicidin (LL-37) concentration | at baseline and every 3 months during supplementation (3,6,9,12 months) up to end of Antarctic residency or 1 year (90-365 days), whichever came first

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Borzutzky, M.D., Principal Investigator — School of Medicine, Pontificia Universidad Católica de Chile

IPD SHARING:
Plan to Share IPD: Undecided